CLINICAL TRIAL: NCT03869086
Title: The Effects of Blueberry Anthocyanin Metabolism on Acute Cardiometabolic Health
Brief Title: Metabolism of Anthocyanins and Heart Health
Acronym: AMP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 related inability to complete study
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: AMP001_22NOV2018
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Blueberry; Metabolism; Anthocyanins; Inter-individual variation; Cardiometabolic health

STUDY DESIGN:
Intervention Model Description: Our research design involves screening individuals and then prospectively recruiting on the basis of two distinct blueberry metabolism profiles based on our previous research findings (in a population with metabolic syndrome). Our study will assess whether individuals with SLOW and FAST anthocyanin metabolism profiles respond differently and will test if the difference in processing may influence cardio metabolic responses. Our study involves feeding a single energy-dense meal which we anticipate will have a transient deleterious effect on acute markers of health. We will test whether adding blueberries to the energy dense meal improves acute responses compared against when adding the equivalent isocaloric amount of placebo. Participants will experience the blueberry and placebo treatments in random order
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomised allocation of treatment order for each participant will be performed by an independent researcher with experience in statistical randomisation. The Principle Investigator will receive notification of the treatment coding order for each subject (in a tamper-evident sealed envelope) which will be prepared by the independent researcher trained in statistics. The coding of the treatment randomisation will only be known to this researcher; and will only be broken at the analysis stage of the study unless a serious adverse event occurs. As the intervention material is a powdered food product, or placebo material, it is considered unlikely that this eventuality may occur.
  During the analysis stage, a blind review of data quality and outlier data will be performed prior to unblinding. Researchers analysing the raw data will remain blind and the data will be locked prior to unblinding of the statistician (which will only occur after the completion of the statistical analysis).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLOW anthocyanin metabolisers (Experimental): Participants will be prospectively recruited to the SLOW anthocyanin metaboliser group, following a pre-intervention screen (blueberry challenge). Participants in this arm will consume (in random order) blueberry and placebo interventions (both consumed with an energy dense meal) in a cross-over manner. At least 7 days washout will be observed between the two treatments.
  Interventions: Other: Freeze dried blueberry powder; Other: Anthocyanin free, sugar-matched placebo
- FAST anthocyanin metabolisers (Experimental): Participants will be prospectively recruited to the FAST anthocyanin metaboliser group, following a pre-intervention screen (blueberry challenge). Participants in this arm will consume (in random order) blueberry and placebo interventions (both consumed with an energy dense meal) in a cross-over manner. At least 7 days washout will be observed between the two treatments.
  Interventions: Other: Freeze dried blueberry powder; Other: Anthocyanin free, sugar-matched placebo

INTERVENTIONS:
Other: Freeze dried blueberry powder — 36 g of freeze-dried blueberry powder to be mixed with milk and served together with an energy-dense meal.
Other: Anthocyanin free, sugar-matched placebo — 36 g of isocaloric placebo, matched for sugars to be mixed with milk and served together with an energy-dense meal.

SUMMARY:
This study aims to find out if consuming a single dose of blueberries, rich in anthocyanins, within an energy dense meal, improves blood vessel function and biomarkers of heart health. The study specifically aims to confirm if differences in how individuals process the bioactive compounds in blueberries, called anthocyanins, has an influence on heart health. The investigators will assess the effects of eating one portion of blueberries on vascular health over a 48hour period, and will track the breakdown compounds within blood and urine, to see if health effects are related to metabolism.

DETAILED DESCRIPTION:
The primary aim of this cross-over designed, placebo controlled, acute dietary intervention study, is to prospectively recruit participants on the basis of anthocyanin metabolism profiles (based on profiles confirmed in our previous studies) following a 'blueberry challenge'. Acute cardio and metabolic function responses will be assessed (by metaboliser profile), following an energy dense test meal with/without the addition of blueberries.

Participants will be healthy, but overweight and obese (BMI inclusion: ≥ 25kg/m2) men and women (aged 50 y to 80 y), who will initially undertake a 'blueberry challenge' by consuming a single dose of freeze dried blueberries. Anthocyanin metaboliser type will be profiled from the analysis of metabolites within urine, collected for 48h following the 'challenge'.

A total of 70 participants will complete the intervention (n=35 FAST and n=35 SLOW metabolisers) which consists of two, test meal periods (separated by at least 7d and allocated in random order); 1) energy dense test meal plus freeze dried blueberries, 2) energy dense test meal plus an isocaloric matched placebo material. Urine samples and ambulatory blood pressure measures will be collected for 24h prior to, and then over the 48h period which follows the test meal intake. Further assessment of vascular and metabolic function will be made at pre-defined times over the 48h postprandial period. Dietary restrictions to abstain from blueberries and reduce the anthocyanin intake level, will be applied for 5d before each test meal intake. In addition, all food and drink will be provided for a 4d period (2d before and during the 48h following the energy dense test meal) to further control the intake of flavonoids and to standardise the influence of background diet on metabolism profile.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 25 kg/m2
* Adults aged 50 - 80 years old
* Successful biochemical, haematological, and urinalysis assessment at screening

Exclusion Criteria:

* Current smokers, or ex-smokers ceasing < 6 months ago
* existing or significant past medical history of vascular disease or medical conditions likely to affect the study measures
* Fructose or lactose intolerant subjects or known allergies to intervention treatments
* Those unprepared to adhere to dietary instructions
* Parallel participation in another research project involving dietary intervention and/or sampling of biological fluids/material
* Those on therapeutic diets or having experienced substantial weight loss within 2 months of screening.
* Those taking flavonoid, nitrate / nitrite containing or fish oil containing supplements (and unwilling to cease intake during, and 1 month preceding the trial) or unwilling to maintain existing intake of other supplements.
* Prescribed hypoglycaemic, anti-hypertensive, vasodilator or hormone replacement therapy (HRT) medication.
* Unsatisfactory biochemical, haematological or urinary results or measurements considered to be counter indicative for the study
* Undiagnosed hypertension (elicited at screening; i.e. ≥ 180 / 110mmHg) at a level requiring immediate referral back to general practitioner for follow-up

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Brachial artery endothelial function | assessed at 0, 1.5, 3, 6, 24, 48 hours after intervention intake
  percentage maximum dilatation assessed via flow mediated dilation (%FMD): (diametermax-diameterbaseline) / diameterbaseline×100.

SECONDARY OUTCOMES:
Office blood pressure | Assessed at 0, 3, 6, 24, 48 hours after intervention intake.
  Measurements of blood pressure
Bioavailability - serum | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of flavonoid and metabolite levels in blood samples
Postprandial Insulin response | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of postprandial insulin control
Total cholesterol | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of blood cholesterol

OTHER OUTCOMES:
Microbiome assessment of phyla and species | Sample collected up to 2 days prior to test meal 1 and assessed within 5 years of study completion
  Assessment of the gut microbiome from faecal samples collected from FAST and SLOW anthocyanin metabolisers.
Ambulatory blood pressure | 1 day before, and the two days following the intake of each energy dense test meal
  Measurement of pre-intervention and postprandial ambulatory blood pressure
Aortic arterial stiffness (cf-PWV) | assessed at 0, 3, 6, 24, 48 hours after intervention intake
  Measurement of carotid to femoral pulse wave velocity
Systemic arterial stiffness (AIx) | assessed at 0, 3, 6, 24, 48 hours after intervention intake
  Measurement of brachial augmentation index (adjusted to 75 beats per minute heart rate)
Bioavailability - urine | 3 days during the blueberry challenge (1 day before and the two days of the assessment) and 3 days during each test meal assessment (1 day before and the two days of the assessment)
  Assessment of flavonoid and metabolite levels in 24 hour urine samples
Postprandial glucose response | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of postprandial glucsoe control
High density lipoprotein cholesterol | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of blood high density lipoprotein cholesterol
Triglycerides | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of blood triglycerides
Low density lipoprotein cholesterol | Measured prior to, and then at +20, +40, +60, +90, +120, +180, +270 and +360 minutes, +24 hours and +48 hours following the energy dense meal intake.
  Assessment of blood low density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Aedin Cassidy, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Quadram Institute Clinical Research Facility; a partnership facility of the NHS, UEA and QIB, Norwich, Norfolk, United Kingdom